CLINICAL TRIAL: NCT01970514
Title: Temporary Axial Rotation Stabilization for Lumbar Disc Prolapse Surgery With the ARO® Spinal System: A Non-randomized Prospective Analysis of Clinical Efficacy, Safety and Cost Effectiveness
Brief Title: Safety Study of ARO Spinal System as an Adjunct to Lumbar Decompression
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ARO Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARO-01
Record Dates: First submitted 2013-10-23; First posted 2013-10-28 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Lumbar Disc Prolapse With Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARO Spinal System (Experimental): ARO Spinal System
  Interventions: Device: ARO Spinal System

INTERVENTIONS:
Device: ARO Spinal System — The device provides an internal axial rotation orthosis (ARO) for patients being surgically treated for herniated nucleus pulposus (HNP).

SUMMARY:
To evaluate the clinical safety and effectiveness of the ARO Spinal System and to assess preliminary cost/benefit analysis in patients undergoing decompression surgery for symptomatic lumbar disc herniations.

The general hypothesis is that the ARO significantly improves outcomes in patients undergoing decompression surgery for symptomatic lumbar disc herniations.

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

1. Radicular pain and evidence of nerve-root irritation lasting 6 weeks or more as evidenced by both:

   1. Radicular pain - below the knee,
   2. Nerve root irritation

   i. positive nerve root tension sign - straight leg raise positive between 30 and 70 degrees, or ii. positive femoral tension sign, or iii. neurologic deficit - asymmetrical depressed reflex or decreased sensation in a dermatomal distribution or weakness in a myotomal distribution.
2. Primary one-level posterolateral herniation in the lower lumbar spine (L4-L5 or L5-S1 only) as shown by magnetic resonance (MR) imaging (protrusion, extrusion or sequestered fragment) consistent with the clinical symptoms (both level and side).
3. The investigator confirms that the patient is a surgical candidate for discectomy,
4. The patient has been scheduled for their surgical procedure no more than two months from time of consent,
5. 18 years to 55 years of age at time of consent,
6. Willing to complete the study requirements and permit agency and sponsor authorized personnel to access medical records,
7. Able to understand oral and written Danish.

Exclusion Criteria:

1. Previous lumbar surgery
2. Cauda equine syndrome
3. Scoliosis greater than 15 degrees
4. Osteoporosis
5. Segmental instability (> 10 degrees angular motion or >4mm translation)
6. Vertebral fractures
7. Spinal Infections
8. Spinal tumors
9. Inflammatory spondyloarthropathy
10. Pregnancy or the intent to become pregnant in the following year
11. Comorbid conditions contraindicating surgery
12. Multiple herniations
13. Known allergy to titanium, aluminum or vanadium
14. Female patients of childbearing age, who are not willing to use adequate contraception specified as: intrauterine devices, hormonal contraceptives (contraceptive pills, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release). It is accepted in certain cases to include subjects having a sterilized permanent partner or subjects using double barrier contraceptive methods which is a condom combined with a diaphragm.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Safety profile compared to historical controls and improvement in leg and back pain | One year

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) improvement is superior to historical control | 1 year
VAS back pain improvement is superior to historical control | 1 year
VAS leg pain improvement is superior to historical control, | 1 year

OTHER OUTCOMES:
The percentage of patients very or somewhat satisfied with their symptoms is greater than historical control | 1 year
There is an increase in the percentage of patients with evidence of annular healing in comparison to historical control | 1 year
There is a decrease in the percentage of patients with evidence of facet degenerative changes in comparison to historical control | 1 year
There is a reduction in the percentage of patients with degenerative changes in the disc in comparison to historical control | 1 year
There is a reduction in the axial rotation motion on the operative level compared to pre-operative motion | 1 year
Surgery with the device has no neurological impact | 1 year
The rate of reherniation is less than in historical control | 1 year
The percent of patients disabled at one year is less than in historical controls | 1 year
The device has a neutral cost/benefit profile in comparison to historical controls to permit further clinical study | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Cody Bunger, MD, DrMedSc, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark